CLINICAL TRIAL: NCT04562623
Title: Prospective Study of Immune Alterations in Operable Breast and Ovarian Carcinoma
Acronym: GYNECO-IMM&CO
Status: Recruiting | Type: Observational
Sponsor: Centre Leon Berard (Other)
Collaborators: Centre de Recherche en Cancérologie de Lyon (CRCL) (Unknown)
Responsible Party: Sponsor
Other Study IDs: ET19-283
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Ovarian Carcinoma; Breast Carcinoma
Keywords: Ovarian cancer; Breast cancer; Immune alterations; Predictive biomarkers
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor samples : FFPE and fresh samples (Fragment of surgery specimen, mastectomy) ; Blood samples (total blood (plasma isolation, circulating DNA, circulating RNA, constitutional DNA and PBMC) and serum)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A : High grade serous ovarian carcinoma
- Cohort B :Breast carcinoma SBR grade II or III: Breast carcinoma SBR grade II or III superior to 3 cm
- Cohort C : Extended Breast carcinoma In situ: Extended Breast carcinoma In situ associated with invasive nodule carcinoma macroscopically visible and eligible to mastectomy

SUMMARY:
GYNECO-IMM&Co is a prospective clinical and biological cohort ; this study aims to identify immune surveillance and escape mechanisms and also predictive biomarkers for survival patients who suffer from ovarian and breast carcinoma.

DETAILED DESCRIPTION:
Breast cancer is the main cancer in women and is the second cause of mortality by cancer in the world for women ; high grade serous ovarian cancer is a rare pathology but survival is less 25% at 5 years.

Breast and ovarian cancers are complex entities with heterogeneous tumor cells but also normal cells including immune cells with represent the microenvironment of the tumor.This microenvironment limits tumor progression but also has been shown to play a crucial role in disease progression, tumor angiogenesis, maintenance and resistance to anticancer therapies.

Despite newly developed immunotherapies, only one-third of patients with breast and ovarian cancer responds to checkpoint inhibitors ; so today there is poor benefit to treat breast and ovarian cancers with immunotherapies. Therefore it needs to better understand immune mechanisms which reduce treatment efficacy. The aim of this clinical study is to better understand mechanisms of immune response inhibition in breast and ovarian cancers. It would characterize actionable targets in patients with resistance to conventional anticancer treatments or immunotherapies.In this context, the hypothesis is that some specific phenotypical or functional alterations of specific immune cells populations (DC, LB, plasmocytes IgA, neutrophils, NK cells, CD8+CD39+ LT, Treg) induce tumoral progression in breast and ovarian cancer. These immune populations will be described (qualitative, quantitative and functional descriptions ; proteic, transcriptomic and genomic profiles) in order to i) determine new immune surveillance mechanisms ii) new targets which allow efficient antitumoral immunity in breast and ovarian cancers.

ELIGIBILITY:
Inclusion Criteria:

* I1. Female patients aged ≥ 18 tears at time of inform consent signature.
* I2. Patient with planned primitive tumor surgery listed below : High grade serous ovarian carcinoma (cohort A), Breast carcinoma SBR grade II or III > 3 cm (cohort B), Extended breast carcinoma In situ associated with invasive nodule carcinoma macroscopically visible and eligible to mastectomy (cohort C).

Note : Patients previously treated by neoadjuvant chemotherapy are eligible and all chemotherapies are authorized.

* I3. Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures and should be willing to comply procedures required per protocol.
* I4. Patient must be covered by a medical insurance.

Exclusion Criteria:

* E1. Patient under guardianship or trusteeship.
* E2. Cancer with constitutional BRCA1/2 mutation.
* E3. Previously treated by immunomodulators (PD1/PDL1, CTLA4).
* E4. Systemic treatment by an immunosuppressor (including, but not limited to, corticosteroids, azathioprine, methotrexate, thalidomide and anti-TNF-alpha) or by an immunostimulant within 2 weeks before inclusion, except corticosteroids listed below: inhaled corticosteroids, intranasal corticosteroids, topic corticosteroids, and systemic corticosteroids with prednisone or equivalent physiological dose ≤ 10 mg/day.
* E5. Patient with known history of autoimmune disease including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis,systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipids syndrome, Wegener syndrome , Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vascularitis, or glomerulonephritis, B or C hepatitis infection, HIV infection.
* E6. Patient with other active tumor except if the tumor is considered not to interfere with outcome measures following sponsor approval such as basal or squamous cell skin cancer. Patient previously treated for an other cancer and without relapse for at least one year are eligible.
* E7. Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients with operable ovarian or breast cancer : patients with high grade serous ovarian carcinoma (cohort A), Breast carcinoma SBR grade II or III > 3 cm (cohort B), Extended breast carcinoma In situ associated with invasive nodule carcinoma macroscopically visible and eligible to mastectomy (cohort C).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Characterization of immune cells populations on tumour sample from exeresis | At surgery
  Frequency, phenotype and function/activation status of immune cells will be determined by flow cytometry, electrochemiluminescence and proliferation test

SECONDARY OUTCOMES:
Characterization of immune cells populations on blood sample | At surgery
  Frequency, phenotype and function/activation status of immune cells will be determined by flow cytometry and electrochemiluminescence
Characterization of transcriptomic profile of immune cells populations | At surgery
  Biomarkers expression, activation or inhibition of functional pathways will be determined by transcriptome sequencing (RNAseq and single cell RNAseq) on tumor sample
Characterization of molecular profile of tumor sample | At surgery
  Genes profile (Mutation, amplification, insertion, deletion) will be determined by whole exome sequencing (WES)
Comparison of soluble factors of the tumor microenvironment with soluble factors present in the blood | At surgery
  Comparative characterization (nature and concentration) by Luminex technology MSD
Characterization of immunoglobulins and their antigenic targets | At surgery
  Characterization by Elisa and Luminex
Characterization of TCR repertory of LT CD8+ and Tregs | At surgery
  TCR repertory of LT CD8+ and Tregs will be determined by transcriptomic profile by RNAseq
Determination of the correlation between biological characterizations at surgery and clinical characterizations | Up to 60 months
  Clinical characterizations are consistent with treatment response and survival ; biological characteristics will describe molecular and transcriptomic profile of the tumor.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Léon Bérard, Lyon, France